CLINICAL TRIAL: NCT00415987
Title: Hematopoietic Stem Cell Transplantation in Myeloma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 572
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Hematopoietic Stem Cell Transplantation

SUMMARY:
The treatment assignment is based on the presence or absence of an HLA-identical sibling donor (Genetic Randomisation, NOT formal Randomisation). Patients with suitable HLA-identical sibling donors are offered a tandem transplant approach consisting of standard autografting nonmyeloablative radiotherapy and allografting. Patients without HLA-identical siblings are treated with standard double autologous transplantation as per Institutional guidelines or enrolled in other treatment programs approved by local IRBs.This is a multi-center study. The Division of Hematology of University of Torino at the S.G.B. Hospital, Torino, Italy, is the co-ordinating Center.

ELIGIBILITY:
Inclusion Criteria:

* Durie-Salmon stage IIA-IIIB multiple myeloma;
* Age > 18 and ≤ 65 years;
* previously untreated myeloma;
* presence of a sibling (potential donor);
* bilirubins < twice normal;ALAT and ASAT < four times normal;
* left ventricular ejection fraction > 40%;
* creatinine clearances > 40 mL/min;
* Pulmonary dysfunction with diffusing capacity for carbon monoxide (DLCO) > 40% and/or need for continuous oxygen supplementation;
* Karnofsky performance status > 60%;
* patients must give written informed consent;

Exclusion Criteria:

* Age > 65 years
* previously treated myeloma;
* absence of a sibling (genetic randomisation cannot be applied);
* Karnofsky performance status score < 60%
* HIV-infection;
* pregnancy;
* Refusal to use contraceptive techniques during and for 12 months following treatment
* patients unable to give written informed consent

PS. Informed consent is obtained from each patient according to the Institutional Review Boards of the participating centers. The study is conducted according to the Declaration of Helsinki.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2006-09

PRIMARY OUTCOMES:
Survival Outcomes

SECONDARY OUTCOMES:
Response Rate
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Bruno, MD, PhD, Principal Investigator — Divisione Ematologia, Università di Torino, Azienda Ospedaliera San Giovanni Battista, Torino, Italy; Mario Boccadoro, MD, Study Director — Divisione Ematologia, Università di Torino, Azienda Ospedaliera San Giovanni Battista, Torino, Italy
Locations (1):
- Ematologia Universitaria Azienda Ospedaliera San Giovanni Battista, Torino, Italy

REFERENCES:
- [Derived] Bruno B, Rotta M, Patriarca F, Mordini N, Allione B, Carnevale-Schianca F, Giaccone L, Sorasio R, Omede P, Baldi I, Bringhen S, Massaia M, Aglietta M, Levis A, Gallamini A, Fanin R, Palumbo A, Storb R, Ciccone G, Boccadoro M. A comparison of allografting with autografting for newly diagnosed myeloma. N Engl J Med. 2007 Mar 15;356(11):1110-20. doi: 10.1056/NEJMoa065464. PMID 17360989